CLINICAL TRIAL: NCT03301935
Title: Risk Assessment in Patients With Symptomatic- and Asymptomatic Preexcitation
Acronym: RASAP
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Jensen-Urstad, Professor, Karolinska University Hospital
Other Study IDs: RASAP
Record Dates: First submitted 2017-02-23; First posted 2017-10-04 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Wolff-Parkinson-White Syndrome
Keywords: Risk assessment
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Electrophysiology testing and exercise stress testing — Each patient will perform an exercise stress test on bicycle before an invasive electrophysiological test. Both examinations will be performed according to current Clinical practice.

SUMMARY:
Prospective cohort study including 150 patients with pre-excitation on ECG referred to our clinic for risk assessment. There will be equal numbers of symptomatic and asymptomatic patients included in the study. Each patient will perform an exercise stress test on bicycle before an invasive electrophysiological test. The purpose of this study is to compare exercise stress testing on bicycle to an invasive electrophysiological study, regarding risk assessment of patients with pre-excitation. The electrophysiology study is set as reference.

DETAILED DESCRIPTION:
Hypothesis:

The sensitivity and specificity for exercise stress test (bicycle) is low in identifying patients with benign accessory pathways and cannot replace an invasive electrophysiological study in risk assessment of symptomatic and asymptomatic patients with pre-excitation. Invasive electrophysiological assessment should be recommended for all patients with pre-excitation despite symptoms or documented arrhythmia.

Methods:

Prospective cohort study including 150 patients with pre-excitation on ECG referred to our clinic for risk assessment. There will be equal numbers of symptomatic and asymptomatic patients included in the study. Each patient will perform an exercise stress test on bicycle before an invasive electrophysiological test. The purpose of this study is to compare exercise stress testing on bicycle to an invasive electrophysiological study, regarding risk assessment of patients with pre-excitation. The electrophysiology study is set as reference.

A. Instruments and methods for analysis:

* All patients will perform an exercise stress test on a test bike according to standard protocol. ECG will be monitored closely regarding loss of pre-excitation during exercise.
* After exercise testing all patients will undergo an invasive electrophysiological study according to standard protocol.

This procedure is set as reference in identifying potentially dangerous accessory pathways.

* APERP as well as shortest R-R interval during atrial fibrillation, when applicable, will be used to characterize the conduction properties of the pathway defining high risk pathway with APERP ≤ 250 ms with or without isoprenaline.
* Inducibility in AVRT (orthodromic or antidromic reentry tachycardia) and atrial fibrillation will be recorded as well as tachycardia cycle length.
* The results of the two tests will be compared with each patient being their own control.

Programmed stimulation for risk assessment in patients with pre-excitation/accessory pathways:

1. AV block or block in AP during IAP, ms
2. VA block or block in AP during IVP, ms
3. Antegrade curve (single ES 600 ms or longer and 400 ms): APERP And AVNERP
4. Retrograde curve (single ES 600 ms): Retrograde APERP and AVNERP
5. Tachycardia induction (Double ES from atrium): Inducibility
6. Burst pacing from atrium
7. Isoprenaline: Dose adjustment until heart rate>100/min or >50% increase from basal level.

   * Antegrade curve during isoprenaline: APERP, AVNERP
   * Retrograde curve during Isoprenaline:

Retrograde APERP and AVNERP

- Tachycardia induction during Isoprenaline

Statistical analysis: Sensitivity, specificity, positive predictive value and negative predictive value of exercise stress test will be assessed, using the electrophysiological study as a reference standard. A true positive and a false negative will be defined, respectively, as the persistence and the disappearance of pre-excitation in the symptomatic and asymptomatic group. A true negative and a false positive will be defined, respectively, as the disappearance and the persistence of pre-excitation in the symptomatic and asymptomatic group. Moreover, we will consider the shortest value between the minimum RR interval during atrial fibrillation and accessory pathway anterograde effective refractory period (APERP) in each patient and look for the value that could be predicted by noninvasive tests with the best combination of sensitivity, specificity, positive and negative predictive value.

Chi Square statistics will be used in comparing categorical data such as inducibility and tachycardia cycle length.

B. Calculation of power: With the planned number of patients, 150, a 10% difference should be detected with a power of 80% at α 0,1.

C. Expected results: We expect exercise testing to have high sensitivity, but low specificity and a low positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular pre exciatation on 12 lead ECG

Exclusion Criteria:

* Inability to perform invasive electrophysiology testing or exercise stress test on bicycle.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with documented ventricular preexcitation, referred for risk assessment to the Arrhythmia department at Karolinska University Hospital, were asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
RASAP | Approximately 1 year from inclusion to 6 months follow-up.
  Number of potentially dangerous pathways (i.e APERP <250 ms) identified by exercise stress test compared to the invasive electrophysiological test in the symptomatic- and asymptomatic Group.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jensen-Urstad, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jemtren A, Saygi S, Akerstrom F, Asaad F, Bourke T, Braunschweig F, Carnlof C, Drca N, Insulander P, Kenneback G, Nordin AP, Sadigh B, Rickenlund A, Saluveer O, Schwieler J, Svennberg E, Tapanainen J, Turkmen Y, Bastani H, Jensen-Urstad M. Risk assessment in patients with symptomatic and asymptomatic pre-excitation. Europace. 2024 Feb 1;26(2):euae036. doi: 10.1093/europace/euae036. PMID 38363996